CLINICAL TRIAL: NCT00825968
Title: Data Collection and Analysis of Patients Who Have Had an Electrophysiological Procedure Performed at the Ross Heart Hospital
Brief Title: Data Collection and Analysis of Patients Who Have Had an Electrophysiological Procedure
Status: Terminated | Type: Observational
Why Stopped: PI stopped study to make a more substantial database.
Sponsor: Emile Daoud (Other)
Responsible Party: Sponsor-Investigator, Emile Daoud, Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2008H0013
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Heart Disease; Atrial Fibrillation
Keywords: Electrophysiological; Heart Disease; Cardiology; Atrial Fibrillation; Risk Factors; Follow-up; Outcomes
MeSH Terms: conditions — Heart Diseases; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Data collection group: Patients having procedures done at the electrophysiology Laboratories at the Ross Heart Hospital at The Ohio State University Medical Center.

SUMMARY:
The purpose of the database is to complete outcomes research of electrophysiological procedures.

DETAILED DESCRIPTION:
The purpose of the database is to complete outcomes research (risk factors, follow-up, procedural data) Perhaps the most important research for any busy clinical laboratory is to appreciate the tendencies and trends that are occurring in their own laboratory setting. This will have a tremendous impact on educating the OSU staff as well as perhaps other centers on best medical practices.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* have or had a procedure preformed in the Electrophysiology Laboratories at the Ross Heart Hospital
* Ability to consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having procedures completed at the electrophysiology Laboratories at the Ross Heart Hospital at The Ohio State University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emile Daoud, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States